CLINICAL TRIAL: NCT04625179
Title: Evaluation of Melatonin and Hyaluronic Acid in Maxillary Sinus Augmentation (a Randomized Controlled Clinical Trial)
Brief Title: Melatonin and Hyaluronic Acid in Maxillary Sinus Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Maxillary sinus augmentation
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy | interventions — Melatonin; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin and hyaluronic acid and sinus membrane elevation (Experimental): melatonin and hyaluronic acid will be placed after maxillary sinus membrane elevation and simultaneous dental implants placement
  Interventions: Other: Melatonin and hyaluronic acid and sinus membrane elevation
- sinus membrane elevation without any materials (Active Comparator): no materials will be placed after maxillary sinus membrane elevation and simultaneous dental implants.
  Interventions: Procedure: sinus membrane elevation without any materials

INTERVENTIONS:
Other: Melatonin and hyaluronic acid and sinus membrane elevation — 3 mg melatonin powder mixed with 0.2% hyaluronic acid gel will be placed to fill the sinus space and around the implant apex.
  Arms: Melatonin and hyaluronic acid and sinus membrane elevation
Procedure: sinus membrane elevation without any materials — No materials will be placed at the sinus space.
  Arms: sinus membrane elevation without any materials

SUMMARY:
melatonin proved an ability to repair bone defects and enhance osseointegration of dental implants. Also, hyaluronic acid has osteopromoting properties.

the effect of melatonin and hyaluronic acid on the newly formed bone in maxillary sinus augmentation was evaluated

DETAILED DESCRIPTION:
16 participants with missing maxillary posterior teeth and residual alveolar ridge of at least 5 mm will be equally and randomly divided into two groups.

The study group will receive melatonin and hyaluronic acid after sinus membrane elevation and simultaneous implant placement while the control group will not receive any materials after sinus membrane elevation and simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Age range will be between (30 - 50) years old.
* Patients with missed one or more of posterior teeth with minimum residual bone height 5 mm
* Adequate inter-occlusal space of at least 8 mm

Exclusion Criteria:

* Maxillary sinus diseases.
* Previous sinus surgery like the Caldwell-Luc operation.
* History of chemotherapy or radiotherapy to maxilla.
* Presence of Underwood's septa/severe sinus floor convolutions.
* Systemic disease affecting bone metabolism.
* Uncontrolled diabetes mellitus.
* Heavy smokers.
* Para functional habits.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
change Implant stability | at baseline and 6 months
  The result is presented as an ISQ value of 1-100. The acceptable stability range lies between 55-85 ISQ. The higher the ISQ, the more stable the implant
change in bone density | at baseline, 1 month and 6 months
  radiographical evaluation using CBCT
change in vertical bone height | at baseline, 1 month and 6 months
  radiographical evaluation using CBCT
change in marginal bone level | at baseline, 1 month and 6 months
  radiographical evaluation using CBCT

SECONDARY OUTCOMES:
Postoperative pain | after 1 week
  based on a 4-point verbal descriptive scale as following: no pain, mild (recognizable but not discomforting pain that required no analgesics), moderate (discomforting but bearable pain and analgesics if used were effective in relieving pain) and severe (difficult to bear and analgesics were effective in relieving pain).
Postoperative swelling | after 1 week
  none (no inflammation), mild (intraoral swelling confined to the surgical field), moderate (extraoral swelling in the surgical zone) and severe (extraoral swelling spreading beyond the surgical zone).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt